CLINICAL TRIAL: NCT00002005
Title: A Phase I Study of Recombinant CD4(rCD4) in Patients With AIDS and AIDS-Related Complex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 064B; CO036g; Serial Number 002
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-01

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; Antigens, CD4; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — CD4 Antigens

INTERVENTIONS:
Drug: CD4 Antigens

SUMMARY:
To determine the safety profile and maximum tolerated dose (MTD) of recombinant soluble human CD4 (rCD4) therapy in patients with AIDS or AIDS related complex (ARC). To obtain a preliminary indication of the antiviral effects of rCD4 in patients with AIDS and ARC. To measure steady state serum levels of rCD4 following continuous infusion therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* Diagnosis of AIDS or AIDS related complex (ARC).
* Failure to tolerate or respond to zidovudine (AZT) or decided to decline AZT therapy.
* The ability to sign a written informed consent form prior to treatment.
* A willingness to abstain from all other experimental therapy for HIV infection during the entire study period.
* A life expectancy of at least 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Serious active opportunistic infections.
* Malignancies other than Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Corticosteroids.
* Nonsteroidal anti-inflammatory agents (NSAI).
* Other experimental therapy.

Patients with the following are excluded:

* Serious active opportunistic infections.
* Malignancies other than Kaposi's sarcoma.

Prior Medication:

Excluded within 3 weeks of study entry:

* Zidovudine (AZT).
* Chemotherapy.
* Immunomodulators.
* Other experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Genentech Inc, South San Francisco, California, United States

REFERENCES:
- [Derived] Arranz R, Garcia-Noblejas A, Grande C, Cannata-Ortiz J, Sanchez JJ, Garcia-Marco JA, Alaez C, Perez-Calvo J, Martinez-Sanchez P, Sanchez-Gonzalez B, Canales MA, Conde E, Martin A, Arranz E, Terol MJ, Salar A, Caballero D. First-line treatment with rituximab-hyperCVAD alternating with rituximab-methotrexate-cytarabine and followed by consolidation with 90Y-ibritumomab-tiuxetan in patients with mantle cell lymphoma. Results of a multicenter, phase 2 pilot trial from the GELTAMO group. Haematologica. 2013 Oct;98(10):1563-70. doi: 10.3324/haematol.2013.088377. Epub 2013 Jun 10. PMID 23753021
- [Derived] Picado A, Singh SP, Rijal S, Sundar S, Ostyn B, Chappuis F, Uranw S, Gidwani K, Khanal B, Rai M, Paudel IS, Das ML, Kumar R, Srivastava P, Dujardin JC, Vanlerberghe V, Andersen EW, Davies CR, Boelaert M. Longlasting insecticidal nets for prevention of Leishmania donovani infection in India and Nepal: paired cluster randomised trial. BMJ. 2010 Dec 29;341:c6760. doi: 10.1136/bmj.c6760. PMID 21190965